CLINICAL TRIAL: NCT02495077
Title: Randomized Controlled Trial of Infliximab (Remicade®) Induction Therapy for Deceased Donor Kidney Transplant Recipients (CTOT-19)
Brief Title: Effects of Inhibiting Early Inflammation in Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT CTOT-19; U01AI063594 (NIH); NIAID CRMS ID#: 20678 (Other: DAIT NIAID)
Record Dates: First submitted 2015-07-06; First posted 2015-07-13 (Estimated); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Kidney Transplant
Keywords: Kidney Transplantation; infliximab; Tissue Donors; Remicade; Induction Therapy; Deceased Donor Kidney Transplant Recipients
MeSH Terms: interventions — Infliximab; Methylprednisolone; Methylprednisolone Hemisuccinate; Mycophenolic Acid; Tacrolimus; thymoglobulin; Acetaminophen; Loratadine; Prednisone; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): rATG is co-administered with anti-TNFa (infliximab/Remicade®) plus maintenance therapy with tacrolimus, a mycophenolic acid derivative (either MMF or enteric coated MPA) and prednisone.
  Interventions: Biological: Infliximab; Drug: Methylprednisolone; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Biological: Thymoglobulin®; Drug: Acetaminophen; Drug: Loratadine; Drug: Prednisone; Drug: Diphenhydramine
- Control (Active Comparator): Rabbit anti-thymocyte globulin (rATG/Thymoglobulin®) plus placebo (Sterile normal saline) induction followed by maintenance therapy with tacrolimus, a mycophenolic acid derivative (either MMF or enteric coated MPA) and prednisone.
  Interventions: Drug: Methylprednisolone; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Biological: Thymoglobulin®; Drug: Acetaminophen; Drug: Loratadine; Biological: Placebo for Infliximab; Drug: Prednisone; Drug: Diphenhydramine

INTERVENTIONS:
Biological: Infliximab — A single dose, of 3mg/kg infusion
  Other Names: Remicade®
  Arms: Experimental
Drug: Methylprednisolone — 500mg will be Initiated just prior to or at the initiation of transplant surgery and prior to Infliximab and thymoglobulin infusion
  Other Names: Solu-Medrol
Drug: Mycophenolate Mofetil — Administered at a target dose of 2000mg daily, as tolerated, until study closure
  Other Names: MMF; CellCept®
Drug: Tacrolimus — Administered at a target dose of 0.1mg/kg BID, post-op, then adjusted to target trough levels of 8-12ng/ml during 1st 3-months post-op and finally adjusted to target trough levels of 5-8ng/ml until study closure
  Other Names: FK-506; FR-900506; Prograf®
Biological: Thymoglobulin® — Administered daily for 5 days with the intention of achieving a total dose of 4.5 to 6.0 mg/kg, as tolerated
  Other Names: Antithymocyte Globulin [Rabbit]; Rabbit ATG
Drug: Acetaminophen — 30 to 60 minutes prior to the start of the infusion
  * Tylenol, 600 to 1000mg by mouth or
  * Suppository form
  Other Names: Tylenol®
Drug: Loratadine — 30 to 60 minutes prior to the start of the infusion
  * Claritin (Loratadine) 10mg by mouth or
  * Benadryl (Diphenhydramine) 25 or 50 mg by mouth
  Other Names: Claritin®
Biological: Placebo for Infliximab — A single dose is volume matched to Infliximab (250mL) infusion
  Arms: Control
Drug: Prednisone — Prednisone will be administered peri-operatively according to center practice. Prednisone should be gradually tapered to no less than 5 mg/day or 10 mg every other day by 3 months post-transplant thereafter until study closure.
Drug: Diphenhydramine — 30 to 60 minutes prior to the start of the infusion
  * Claritin (Loratadine) 10mg by mouth or
  * Benadryl (Diphenhydramine) 25 or 50 mg by mouth
  Other Names: Benadryl

SUMMARY:
During transplant surgery, there is a period of time when a donated kidney is removed from a donor's body and stored until the time of the transplant surgery. The storage procedure results in buildup of various proteins within the kidney that can injure the donated kidney after it is transplanted. One of these proteins is tumor necrosis factor-alpha (TNF-alpha).

The purpose of this study is to evaluate whether taking infliximab, which blocks tumor necrosis factor alpha (TNF-alpha), just prior to transplant surgery, along with usual transplant medicines will protect the donated kidney from damage caused by TNF-alpha and help keep the transplanted kidney healthy for a longer period of time.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double blind (masked), placebo-controlled, 2-arm clinical trial of 300 deceased donor kidney transplant recipients. Participants will be randomized (1:1) to the experimental or control arm (150 subjects per arm).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years of age) male and female recipients (all races and ethnicities)
2. Subject must be able to understand and provide consent
3. Recipients of deceased donor kidney transplants (including re-transplants)
4. Negative crossmatch, actual or virtual, or a PRA of 0% on historic and current sera as determined by each participating study center
5. Donor kidneys from deceased donors and donors after cardiac death (DCD) with Kidney Donor Profile Indices (KDPI) ranging from ≥20 to <95
6. Female participants of childbearing potential must have a negative pregnancy test upon study entry
7. Subjects must have a negative test result for latent tuberculosis (TB) infection (PPD, QuantiFERON, ELISPOT):

   * Subjects who have a negative test result for latent TB infection within 1 year of transplant date are eligible for enrollment and no further action is required
   * Subjects who have a negative test for latent TB infection that is greater than 1 year old are eligible for enrollment but are required to have a repeat test prior to transplantation.

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Recipients of living donor transplants
3. Presence of other transplanted solid organ (heart, lung, liver, pancreas, small intestines) or co-transplanted organ
4. Human immunodeficiency virus positive (HIV+) recipients
5. Epstein-Barr virus Immunoglobulin G (EBV IgG) negative recipients
6. Hepatitis B surface antigen positive kidney transplant recipients
7. Hepatitis B core antibody positive kidney transplant recipients
8. Hepatitis B negative kidney transplant recipients that receive transplants from Hepatitis B core antibody positive donor
9. Hepatitis C Virus positive (HCV+) patients who are either untreated or have failed to demonstrate sustained viral remission for more than 12 months after anti-viral treatment
10. Recipients with a previous history of active TB
11. Recipients with a positive test for latent TB infection (PPD, QuantiFERON, ELISPOT), regardless of previous therapy
12. Any severe infection at the time of transplantation.

    --Note: Severe infection determination will be made by the local site investigator.
13. Severe congestive heart failure (NYHA functional class III or higher)
14. Subjects with a known hypersensitivity to any murine/ mouse proteins
15. Subjects with any history of receiving any anti-tumor necrosis factor (anti- TNF) products
16. Subjects in whom rabbit anti-thymocyte globulin (Thymoglobulin®) or infliximab might not be tolerated
17. Subjects with a white blood cell count less than 3000/mm^3
18. Subjects with a platelet count less than 100,000/mm^3
19. Subjects with systolic blood pressure <100 mm/Hg
20. Subjects with symptomatic orthostatic hypotension or currently requiring Midodrine for blood pressure support
21. Subjects from, or who have traveled, to endemic areas with a history of active histoplasmosis or, with a chest x-ray consistent with previous active histoplasmosis (no serological testing required) :

    --Endemic regions determined by site based on local standard of care.
22. Subjects currently or formerly residing in regions of the United States that are highly endemic for coccidioidomycosis, and who have a positive serologic test for coccidioidomycosis:

    --Endemic regions determined by site based on local standard of care.
23. Recipients are excluded if the local site decides to treat the recipient with fluconazole because of diagnosis or suspicion of fungal infection the donor
24. Subjects that receive IVIG treatment within 3 months of transplant or planned intravenous immunoglobulin (IVIG) treatment peri-transplant
25. Use of an investigational agent within 4-weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S. Heeger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai, Recanati Miller Transplant Institute; Donald E Hricik, MD, Study Chair — University Hospitals of Cleveland, Division of Nephrology & Hypertension
Locations (15):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - University of Manitoba, Winnipeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Hricik DE, Armstrong B, Alhamad T, Brennan DC, Bromberg JS, Bunnapradist S, Chandran S, Fairchild RL, Foley DP, Formica R, Gibson IW, Kesler K, Kim SJ, Mannon RB, Menon MC, Newell KA, Nickerson P, Odim J, Poggio ED, Sung R, Shapiro R, Tinckam K, Vincenti F, Heeger PS. Infliximab Induction Lacks Efficacy and Increases BK Virus Infection in Deceased Donor Kidney Transplant Recipients: Results of the CTOT-19 Trial. J Am Soc Nephrol. 2023 Jan 1;34(1):145-159. doi: 10.1681/ASN.2022040454. Epub 2022 Oct 4. PMID 36195441
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen sites consented 290 participants for evaluation of eligibility criteria. 242 participants were determined to be eligible and enrolled into this trial.
Pre-assignment Details: 290 potential participants signed an informed consent before undergoing any study procedures. After the informed consent was signed and the participant was determined to meet entry criteria, the participant was enrolled in the study. A total of 242 were determined eligible to start the study.
Groups:
- Experimental: The experimental group underwent a transplant procedure and received rabbit anti-thymocyte globulin (rATG, Thymoglobulin) co-administered with anti-TNFa (infliximab/Remicade®) followed by maintenance therapy with tacrolimus, either Mycophenolate Mofetil/MMF or Mycophenolate Acid/MPA (or their generic equivalents) and prednisone
- Control: The control group underwent a transplant procedure and received rabbit anti-thymocyte globulin (rATG, Thymoglobulin) plus placebo (sterile normal saline) induction followed by maintenance therapy with tacrolimus, either Mycophenolate Mofetil/MMF or Mycophenolate Acid/MPA (or their generic equivalents) and prednisone
- Enrolled, Discontinued Pre-Transplant: Participants who were eligible and enrolled but withdrew from the study prior to receiving a transplant.
- Screen Failure: Participants who were consented but did not meet inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Experimental | Control | Enrolled, Discontinued Pre-Transplant | Screen Failure
Started | 113 | 112 | 17 | 48
Completed | 93 | 91 | 0 | 0
Not Completed | 20 | 21 | 17 | 48
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Death | 3 | 5 | 0 | 0
Not completed — Lost to Follow-up | 6 | 4 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 4 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 48
Not completed — Withdrawal by Subject | 7 | 7 | 7 | 0
Not completed — Covid-19 research restrictions | 1 | 0 | 0 | 0
Not completed — Visit 14 scheduling difficulties | 1 | 0 | 0 | 0
Not completed — Incarcerated | 0 | 1 | 0 | 0
Not completed — Transplant nephrectomy, patient decision | 0 | 1 | 0 | 0
Not completed — Timing of transplant and randomization | 0 | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 113 | 112 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 96 | 189
  >=65 years | 20 | 16 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (10.70) | 53.6 (10.69) | 53.4 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 90
  Male | 71 | 64 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 12 | 29
  Not Hispanic or Latino | 96 | 99 | 195
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 40 | 46 | 86
  White | 51 | 48 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 9 | 21
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 4
  United States | 111 | 110 | 221
Reason for Transplant [Count of Participants; unit: Participants] — The reason for transplant captures a participant's reason/cause of end stage renal disease and their need for transplant.
  Participants
    Diabetes | 28 | 32 | 60
    Glomerular disease | 21 | 18 | 39
    Hypertension | 24 | 23 | 47
    Polycystic kidney disease | 15 | 10 | 25
    Other | 25 | 29 | 54
Donor Cause of Death [Count of Participants; unit: Participants] — Donor cause of death was classified as resulting from a cerebrovascular accident (CVA) or a non-cerebrovascular accident (non-CVA).
  Participants
    CVA | 34 | 22 | 56
    Non-CVA | 79 | 90 | 169

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between the Mean eGFR (Modified MDRD) in the Experimental vs. Control Groups.
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Modification of Diet in Renal Disease (MDRD) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. eGFR values from months 1, 3, 6, 12, 18, and 24 were used to generate an estimate of the month 24 eGFR for each treatment group.
Time Frame: 24-Month post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available eGFR data.
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 111 | 109
mL/min/1.73m2 | 52.45 [48.38 to 56.52] | 57.35 [53.18 to 61.52]
Statistical Analysis 1: Comparison: Experimental vs Control; Mean eGFR of the two treatment groups was compared. The p-value, estimated month 24 eGFR within each treatment group, estimate of the treatment group difference, and estimated 95% confidence intervals result from a repeated measures mixed model using available eGFR data from months 1, 3, 6, 12, 18, and 24 to compare the experimental group to the control group. Random effects for the intercept and eGFR collection day were utilized in the model; Test type: Superiority; p = 0.099, Mixed Models Analysis; Mean Difference (Final Values) = -4.90, 95% CI 2-sided [-10.73 to 0.93]

2. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Cellular Rejection (BPAR)
Description: Acute cellular rejection was defined based on central lab pathology interpretation using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to IA with or without clinical symptoms within 6 months of transplant were determined to have met the endpoint. Severity is graded as IA, IB, IIA, IIB, or III, with IA being the mildest form of cellular rejection and III being the most severe form of cellular rejection.Criteria include: IA-significant interstitial infiltration and foci of moderate tubulitis; IB-significant interstitial infiltration and foci of severe tubulitis; IIA-mild to moderate intimal arteritis; IIB-severe intimal arteritis; III-transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation.
Time Frame: 6 month post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available central pathology read data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 71 | 66
percentage of participants | 4.2 [0.9 to 11.9] | 3.0 [0.4 to 10.5]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p > 0.999, Fisher Exact

3. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Cellular Rejection (BPAR).
Description: Acute cellular rejection was defined based on central lab pathology interpretation using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to IA with or without clinical symptoms within 24 months of transplant were determined to have met the endpoint. Severity is graded as IA, IB, IIA, IIB, or III, with IA being the mildest form of cellular rejection and III being the most severe form of cellular rejection. Criteria include: IA-significant interstitial infiltration and foci of moderate tubulitis; IB-significant interstitial infiltration and foci of severe tubulitis; IIA-mild to moderate intimal arteritis; IIB-severe intimal arteritis; III-transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation.
Time Frame: 24 months post-transplantation
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 71
percentage of participants | 5.1 [1.4 to 12.6] | 4.2 [0.9 to 11.9]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p > 0.999, Fisher Exact

4. Secondary Outcome: BANFF Grades of First Acute Cellular Rejections (ACR).
Description: as for outcome 2
Time Frame: 6 month post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants who had ACR within the first 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 3 | 2
Participants
  IA | 1 | 1
  IB | 1 | 0
  IIA | 1 | 1
  IIB | 0 | 0
  III | 0 | 0

5. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Cellular Rejection (BPAR) or Borderline Rejection.
Description: Acute cellular rejection was defined based on central lab pathology interpretation using the Banff 2007 criteria. Participants with a Banff grade of borderline or greater than or equal to IA with or without clinical symptoms within 6 months of transplant were determined to have met the endpoint. Severity is graded as Borderline, IA, IB, IIA, IIB, or III, with borderline representing possible cellular rejection, IA being the mildest form of cellular rejection, and III being the most severe form of cellular rejection.Criteria include: Borderline-no intimal arteritis is present but foci of mild tubulitis; IA-significant interstitial infiltration and foci of moderate tubulitis; IB-significant interstitial infiltration and foci of severe tubulitis; IIA-mild to moderate intimal arteritis; IIB-severe intimal arteritis; III-transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation.
Time Frame: 6 months post-transplantation
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 71 | 66
percentage of participants | 8.5 [3.2 to 17.5] | 6.1 [1.7 to 14.8]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.746, Fisher Exact

6. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Cellular Rejection (BPAR) or Borderline Rejection
Description: Acute cellular rejection was defined based on central lab pathology interpretation using the Banff 2007 criteria. Participants with a Banff grade of borderline or greater than or equal to IA with or without clinical symptoms within 24 months of transplant were determined to have met the endpoint. Severity is graded as Borderline, IA, IB, IIA, IIB, or III, with borderline representing possible cellular rejection, IA being the mildest form of cellular rejection, and III being the most severe form of cellular rejection. Criteria include: Borderline-no intimal arteritis is present but foci of mild tubulitis; IA-significant interstitial infiltration and foci of moderate tubulitis; IB-significant interstitial infiltration and foci of severe tubulitis; IIA-mild to moderate intimal arteritis; IIB-severe intimal arteritis; III-transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation.
Time Frame: 24 months post-transplantation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 71
percentage of participants | 12.8 [6.3 to 22.3] | 7 [2.3 to 15.7]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.242, Chi-squared

7. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Antibody Mediated Rejection (AMR)
Description: Antibody mediated rejection (AMR) was defined based on central lab pathology interpretation using the Banff 2013 criteria. Participants with a Banff finding of AMR within 6 months of transplant were determined to have met the endpoint. AMR is classified as acute/active, chronic/active, or C4d staining positive.Criteria include: acute/active-histologic evidence of acute tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of donor-specific antibodies (DSAs); chronic/active-morphologic evidence of chronic tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of DSAs; C4d staining positive-linear C4d staining in peritubular capillaries, glomerulitis=0, peritubular capillary=0, chronic glomerulopathy=0, no acute cell-mediated rejection or borderline changes.
Time Frame: 6 months post-transplantation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 71 | 66
Participants | 0.0 | 0.0

8. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Antibody Mediated Rejection (AMR).
Description: Antibody mediated rejection (AMR) was defined based on central lab pathology interpretation using the Banff 2013 criteria. Participants with a Banff finding of AMR within 24 months of transplant were determined to have met the endpoint. AMR is classified as acute/active, chronic/active, or C4d staining positive. Criteria include: acute/active-histologic evidence of acute tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of donor-specific antibodies (DSAs); chronic/active-morphologic evidence of chronic tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of DSAs; C4d staining positive-linear C4d staining in peritubular capillaries, glomerulitis=0, peritubular capillary=0, chronic glomerulopathy=0, no acute cell-mediated rejection or borderline changes.
Time Frame: 24 months post-transplantation
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 71
percentage of participant | 1.3 [0.0 to 6.9] | 0.0 [NA to NA] — Confidence limits not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p > 0.999, Fisher Exact

9. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Antibody Mediated Rejection AMR or Suspicious for AMR
Description: Antibody mediated rejection (AMR) was defined based on central lab pathology interpretation using the Banff 2013 criteria. Participants with a Banff finding of AMR or suspicious for AMR within 6 months of transplant were determined to have met the endpoint. AMR is classified as acute/active, chronic/active, C4d staining positive, or suspicious. Criteria include: acute/active-histologic evidence of acute tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of donor-specific antibodies (DSAs); chronic/active-morphologic evidence of chronic tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of DSAs; C4d staining positive-linear C4d staining in peritubular capillaries, glomerulitis=0, peritubular capillary=0, chronic glomerulopathy=0, no acute cell-mediated rejection or borderline changes; suspicious-when 2 of 3 factors for acute/active are present.
Time Frame: 6 months post-transplantation
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 71 | 66
percentage of participants | 2.8 [0.3 to 9.8] | 0.0 [NA to NA] — Confidence limits not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.497, Fisher Exact

10. Secondary Outcome: Percent of Participants With Biopsy Proven Acute Antibody Mediated Rejection AMR or Suspicious for AMR.
Description: Antibody mediated rejection (AMR) was defined based on central lab pathology interpretation using the Banff 2013 criteria. Participants with a Banff finding of AMR or suspicious for AMR within 24 months of transplant were determined to have met the endpoint. AMR is classified as acute/active, chronic/active, C4d staining positive, or suspicious. Criteria include: acute/active-histologic evidence of acute tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of donor-specific antibodies (DSAs); chronic/active-morphologic evidence of chronic tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of DSAs; C4d staining positive-linear C4d staining in peritubular capillaries, glomerulitis=0, peritubular capillary=0, chronic glomerulopathy=0, no acute cell-mediated rejection or borderline changes; suspicious-when 2 of 3 factors for acute/active are present
Time Frame: 24 months post-transplantation
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 71
percentage of participants | 3.8 [0.8 to 10.8] | 1.4 [0.0 to 7.6]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.622, Fisher Exact

11. Secondary Outcome: BANFF Grades of First AMR.
Description: Antibody mediated rejection (AMR) was defined based on central lab pathology interpretation using the Banff 2013 criteria. Participants with a Banff finding of AMR within 6 months of transplant were determined to have met the endpoint. AMR is classified as acute/active, chronic/active, or C4d staining positive. Criteria include: acute/active-histologic evidence of acute tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of donor-specific antibodies (DSAs); chronic/active-morphologic evidence of chronic tissue injury, evidence of current/recent antibody interaction with vascular endothelium, and serologic evidence of DSAs; C4d staining positive-linear C4d staining in peritubular capillaries, glomerulitis=0, peritubular capillary=0, chronic glomerulopathy=0, no acute cell-mediated rejection or borderline changes.
Time Frame: 6 months post-transplantation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 71 | 66
Participants | 0 | 0

12. Secondary Outcome: Percent of Participants With BANFF Chronicity Scores > or Equal 2 on the 24 Month Biopsy.
Description: The Banff 2013 classification involves scoring numerous characteristics of renal biopsy specimens. The ci (interstitial fibrosis) and ct (tubular atrophy) scores are two such characteristics. The scores can take values of 0, 1, 2, or 3 for each characteristic (ci and ct), indicating increasing severity of disease as the scores increase. Participants are considered to have met this endpoint if their ci + ct score on the 24 month biopsy summed to be > or equal to 2.
Time Frame: 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available 24 month central pathology read data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 26 | 22
percentage of participants | 73.1 [52.2 to 88.4] | 36.4 [17.2 to 59.3]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.011, Chi-squared

13. Secondary Outcome: Change in BANFF Chronicity Scores Between Implantation and the 24 Month Biopsy.
Description: The Banff 2013 classification involves scoring numerous characteristics of renal biopsy specimens. The ci (interstitial fibrosis) and ct (tubular atrophy) scores are two such characteristics. The scores can take values of 0, 1, 2, or 3 for each characteristic (ci and ct), indicating increasing severity of disease as the scores increase. For this endpoint, the sum of ci+ct scores from the implantation biopsy was subtracted from the sum of the ci+ct scores from the month 24 biopsy and the difference between the two time points was classified as 0, 1, 2, or 3+. Higher values of this difference indicate more severe disease.
Time Frame: 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available ci and ct scores from central pathology on both the implantation and 24 month biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 26 | 18
Participants
  0 | 4 | 6
  1 | 6 | 6
  2 | 9 | 2
  3+ | 7 | 4
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.135, Cochran-Mantel-Haenszel

14. Secondary Outcome: Percent of Participants With Locally Treated Rejection, Defined as Treatment Administered for Rejection Based on Clinical Signs or Biopsy Findings.
Description: Biopsies were read by the local pathologist at the hospital where the participant was a patient. These local reads informed clinical care for the participant, which may or may not include prescribing/administering medication to the participant to help with clinical concerns or findings noted on a biopsy. Participants were considered to have met this endpoint if they have a report of receiving treatment for clinical or biopsy-proven rejection during the first 6 months post-transplant.
Time Frame: 6 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available local pathology read data during the first 6 months of post-transplant follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 95 | 83
percentage of participants | 12.6 [6.7 to 21.0] | 20.5 [12.4 to 30.8]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.157, Chi-squared

15. Secondary Outcome: Percent of Participants With Locally Treated Rejection, Defined as Treatment Administered for Rejection Based on Clinical Signs or Biopsy Findings.
Description: Biopsies were read by the local pathologist at the hospital where the participant was a patient. These local reads informed clinical care for the participant, which may or may not include prescribing/administering medication to the participant to help with clinical concerns or findings noted on a biopsy. Participants were considered to have met this endpoint if they have a report of receiving treatment for clinical or biopsy-proven rejection during the 24 month post-transplant follow-up.
Time Frame: 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available local pathology read data during the 24 month post-transplant follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 99 | 89
percentage of participants | 16.2 [9.5 to 24.9] | 27 [18.1 to 37.4]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.071, Chi-squared

16. Secondary Outcome: Change in eGFR Between 3 Months and 24 Months as Measured by MDRD
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Modification of Diet in Renal Disease (MDRD) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. The change in eGFR between months 3 and 24 was calculated as the month 24 eGFR minus the month 3 eGFR for each participant. A window of +/- 14 days was used for month 3 and +/- 1 month was used for month 24.
Time Frame: 3 months and 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available eGFR data within window at months 3 and 24.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 38 | 41
mL/min/1.73m2 | 2.8 (15.06) | 4.8 (13.26)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.543, t-test, 2 sided

17. Secondary Outcome: Change in eGFR Between 3 Months and 24 Months as Measured by CKD-EPI
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. The change in eGFR between months 3 and 24 was calculated as the month 24 eGFR minus the month 3 eGFR for each participant. A window of +/- 14 days was used for month 3 and +/- 1 month was used for month 24.
Time Frame: 3 months and 24 months post-transplantation
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 38 | 41
mL/min/1.73m2 | 2.7 (16.38) | 4.4 (13.91)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.617, t-test, 2 sided

18. Secondary Outcome: Change in eGFR Between Post-transplant Nadir and 24 Months as Measured by MDRD
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Modification of Diet in Renal Disease (MDRD) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. Post-transplant nadir was defined as the lowest value of eGFR from the first 6 months post-transplant. The change in eGFR between nadir and month 24 was calculated as the month 24 eGFR minus the nadir eGFR for each participant. A window of +/- 21 days was used for month 6 and +/- 1 month was used for month 24.
Time Frame: 6 months and 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available eGFR data within window at months 6 and 24.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 42 | 42
mL/min/1.73m2 | 8.1 (14.06) | 11.6 (14.69)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.275, t-test, 2 sided

19. Secondary Outcome: Change in eGFR Between Post-transplant Nadir and 24 Months as Measured by CKD-EPI
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. Post-transplant nadir was defined as the lowest value of eGFR from the first 6 months post-transplant. The change in eGFR between nadir and month 24 was calculated as the month 24 eGFR minus the nadir eGFR for each participant. A window of +/- 21 days was used for month 6 and +/- 1 month was used for month 24.
Time Frame: 6 months and 24 months post-transplantation
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 42 | 42
mL/min/1.73m2 | 8.5 (15.21) | 12.0 (15.36)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.300, t-test, 2 sided

20. Secondary Outcome: Change in eGFR Between 6 Months and 24 Months as Measured by MDRD
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Modification of Diet in Renal Disease (MDRD) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. The change in eGFR between months 6 and 24 was calculated as the month 24 eGFR minus the month 6 eGFR for each participant. A window of +/- 21 days was used for month 6 and +/- 1 month was used for month 24.
Time Frame: 6 months and 24 months post-transplantation
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 39 | 36
mL/min/1.73m2 | 1.0 (11.73) | 5.2 (13.05)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.152, t-test, 2 sided

21. Secondary Outcome: Change in eGFR Between 6 Months and 24 Months as Measured by CKD-EPI
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. The change in eGFR between months 6 and 24 was calculated as the month 24 eGFR minus the month 6 eGFR for each participant. A window of +/- 21 days was used for month 6 and +/- 1 month was used for month 24.
Time Frame: 6 months and 24 months post-transplantation
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 39 | 36
mL/min/1.73m2 | 0.8 (12.67) | 4.8 (13.42)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.181, t-test, 2 sided

22. Secondary Outcome: eGFR Values as Measured by MDRD
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Modification of Diet in Renal Disease (MDRD) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. eGFR values from day 7 and months 1, 3, 6, 12, 18, and 24 were used to generate an estimate of the eGFR at each time point of interest for each treatment group.
Time Frame: Day 7 post-transplantation
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 112 | 110
mL/min/1.73m2 | 38.93 [35.88 to 41.97] | 39.96 [36.88 to 43.04]
Statistical Analysis 1: Comparison: Experimental vs Control; Day 7. Mean eGFR of the two treatment groups was compared. The p-value, estimated day 7 eGFR within each treatment group, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available eGFR data from day 7 and months 1, 3, 6, 12, 18, and 24 to compare the experimental group to the control group at day 7. Random effects for the intercept and eGFR collection day were utilized in the model; Test type: Superiority; p = 0.639, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-5.37 to 3.30]

23. Secondary Outcome: eGFR Values as Measured by MDRD
Description: as for outcome 22
Time Frame: Days 30, 60, and 180 post-transplantation
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 111 | 109
mL/min/1.73m2
  Day 30 | 46.64 [43.36 to 49.92] | 48.20 [44.89 to 51.51]
  Day 90 | 47.14 [43.90 to 50.38] | 48.99 [45.71 to 52.26]
  Day 180 | 47.89 [44.66 to 51.11] | 50.16 [46.90 to 53.42]
Statistical Analysis 1: Comparison: Experimental vs Control; Day 30. Mean eGFR of the two treatment groups was compared. The p-value, estimated day 30 eGFR within each treatment group, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available eGFR data from months 1, 3, 6, 12, 18, and 24 to compare the experimental group to the control group at day 30. Random effects for the intercept and eGFR collection day were utilized in the model; Test type: Superiority; p = 0.510, Mixed Models Analysis; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-6.22 to 3.10]
Statistical Analysis 2: Comparison: Experimental vs Control; Day 90. Mean eGFR of the two treatment groups was compared. The p-value, estimated day 90 eGFR within each treatment group, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available eGFR data from months 1, 3, 6, 12, 18, and 24 to compare the experimental group to the control group at day 90. Random effects for the intercept and eGFR collection day were utilized in the model; Test type: Superiority; p = 0.430, Mixed Models Analysis; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-6.45 to 2.76]
Statistical Analysis 3: Comparison: Experimental vs Control; Day 180. Mean eGFR of the two treatment groups was compared. The p-value, estimated day 180 eGFR within each treatment group, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available eGFR data from months 1, 3, 6, 12, 18, and 24 to compare the experimental group to the control group at day 180. Random effects for the intercept and eGFR collection day were utilized in the model; Test type: Superiority; p = 0.328, Mixed Models Analysis; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-6.86 to 2.31]

24. Secondary Outcome: eGFR Values as Measured by CKD-EPI
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicates moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or endstage kidney failure. eGFR values from day 7 and months 1, 3, 6, 12, 18, and 24 were used to generate an estimate of the eGFR at each time point of interest for each treatment group.
Time Frame: Day 7 post-transplantation
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 112 | 110
mL/min/1.73m2 | 41.01 [37.68 to 44.33] | 41.85 [38.49 to 45.22]
Statistical Analysis 1: Comparison: Experimental vs Control; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.725, Mixed Models Analysis; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-5.58 to 3.89]

25. Secondary Outcome: eGFR Values as Measured by CKD-EPI
Description: as for outcome 24
Time Frame: Days 30, 90, and 180 post-transplantation
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Experimental | Control
Number analyzed (Participants) | 111 | 109
mL/min/1.73m2
  Day 30 | 49.29 [45.72 to 52.85] | 50.63 [47.03 to 54.24]
  Day 90 | 49.80 [46.27 to 53.32] | 51.44 [47.87 to 55.00]
  Day 180 | 50.56 [47.05 to 54.07] | 52.65 [49.09 to 56.20]
Statistical Analysis 1: Comparison: Experimental vs Control; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p = 0.601, Mixed Models Analysis; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-6.41 to 3.72]
Statistical Analysis 2: Comparison: Experimental vs Control; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.519, Mixed Models Analysis; Mean Difference (Final Values) = -1.64, 95% CI 2-sided [-6.66 to 3.37]
Statistical Analysis 3: Comparison: Experimental vs Control; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.411, Mixed Models Analysis; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-7.08 to 2.91]

26. Secondary Outcome: Percent of Participants With Death or Graft Failure.
Description: Participants who died or experienced graft failure were considered to have met this endpoint. Graft failure was defined as the need for post-transplant dialysis for more than 56 days.
Time Frame: 24 months post-transplantation
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 113 | 112
percentage of participants | 5.3 [2.0 to 11.2] | 7.1 [3.1 to 13.6]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.569, Chi-squared

27. Secondary Outcome: Percent of Participants With Only Graft Failure.
Description: Participants who experienced graft failure were considered to have met this endpoint. Graft failure was defined as the need for post-transplant dialysis for more than 56 days.
Time Frame: 24 months post-transplantation
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 113 | 112
percentage of participants | 2.7 [0.6 to 7.6] | 2.7 [0.6 to 7.6]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p > 0.999, Fisher Exact

28. Secondary Outcome: Percent of Participants That Required at Least One Dialysis Treatment.
Description: Dialysis within the first week post-transplant is used in the setting of delayed graft function (DGF). Participants are considered to have had DGF if they had at least one dialysis treatment in the first week post-transplant.
Time Frame: 1 week post-transplantation
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 113 | 112
percentage of participants | 31.0 [22.6 to 40.4] | 35.7 [26.9 to 45.3]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.451, Chi-squared

29. Secondary Outcome: Number of Dialysis Sessions.
Description: The number of dialysis sessions a person had during their first 8 weeks post-transplant was used for this endpoint.
Time Frame: 8 weeks post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available data during the first 8 weeks.
Measure: Mean (Standard Deviation); unit: Dialysis sessions
Arm/Group | Experimental | Control
Number analyzed (Participants) | 111 | 109
Dialysis sessions | 0.14 (1.0) | 0.26 (2.32)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.614, t-test, 2 sided

30. Secondary Outcome: Duration of Delayed Graft Function (DGF), Defined as Time From Transplantation to the Last Required Dialysis Treatment.
Description: Participants are considered to have had DGF if they had at least one dialysis treatment in the first week post-transplant. For this endpoint, duration was calculated as the date of last post-transplant dialysis treatment minus the date of the first post-transplant dialysis treatment.
Time Frame: First post-transplant dialysis treatment to last post-transplant dialysis treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental | Control
Number analyzed (Participants) | 33 | 39
Days | 13.27 (13.89) | 15.74 (38.37)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.710, t-test, 2 sided

31. Secondary Outcome: Percent of Participants With Primary Non-Function (PNF), Defined as Dialysis-dependency for More Than 3 Months.
Description: Post-transplant dialysis is sometimes required in the setting of kidney transplant. If such dialysis continues for more than 3 months, the participant is considered to have PNF and, as such, meets this endpoint definition.
Time Frame: Transplantation through at least month 3 up to month 24
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available data for dialysis used.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 109 | 107
Percent of Participants | 2.8 [0.6 to 7.8] | 0.9 [0.0 to 5.1]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.622, Fisher Exact

32. Secondary Outcome: Change From Baseline (Immediately After Surgery) in Serum Creatinine.
Description: Serum creatinine (mg/dL) is used to measure kidney function. A normal result is 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women. Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys. eGFR values from 24, 48, and 72 hours post-transplant (i.e., days 1, 2, and 3) were used to generate an estimate of the serum creatinine at each time point of interest for each treatment group.
Time Frame: 24, 48 and 72 hours post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available serum creatinine data during the first 72 hours post-transplant.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Experimental | Control
Number analyzed (Participants) | 113 | 111
mg/dL
  24 Hours | 7.35 [6.74 to 7.95] | 6.85 [6.24 to 7.46]
  48 Hours | 6.24 [5.64 to 6.84] | 5.87 [5.26 to 6.48]
  72 Hours | 5.77 [5.16 to 6.37] | 5.21 [4.60 to 5.81]
Statistical Analysis 1: Comparison: Experimental vs Control; 24 Hours/Day 1. Mean serum creatinine of the two treatment groups was compared. The p-value, estimated 24 hour creatinine level within each treatment group, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available serum creatinine data from 24, 48, and 72 hours to compare the experimental group to the control group at 24 hours/day 1. A random effect for the intercept was utilized in the model; Test type: Superiority; p = 0.256, Mixed Models Analysis; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.36 to 1.35]
Statistical Analysis 2: Comparison: Experimental vs Control; 48 Hours/Day 2. Mean serum creatinine of the two treatment groups was compared. The p-value, estimated 48 hour creatinine level within each treatment group, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available serum creatinine data from 24, 48, and 72 hours to compare the experimental group to the control group at 48 hours/day 2. A random effect for the intercept was utilized in the model; Test type: Superiority; p = 0.391, Mixed Models Analysis; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.48 to 1.23]
Statistical Analysis 3: Comparison: Experimental vs Control; 72 Hours/Day 3. Mean serum creatinine of the two treatment groups was compared. The p-value, estimated 72 hour creatinine level within each treatment group, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available serum creatinine data from 24, 48, and 72 hours to compare the experimental group to the control group at 72 hours/day 3. A random effect for the intercept was utilized in the model; Test type: Superiority; p = 0.199, Mixed Models Analysis; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-0.30 to 1.42]

33. Secondary Outcome: Days From Transplantation Until Event (ACR, AMR, or Hospitalization for Infection and/or Malignancy)
Description: Participants are considered to have met this endpoint if they experienced biopsy-proven T-cell mediated rejection (ACR) or antibody mediated rejection (AMR) based on central pathology reading or were hospitalized for infection and/or malignancy. For participants who met one or more of these three components, the earliest event date of the three components was used as the time of meeting the endpoint. Participants who did not meet any of the three components were censored at their last date of follow-up. Event (or censor) day was calculated as event (or censor) date minus transplant date.
Time Frame: 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants with available central pathology data and hospitalization data.
Measure: Median (95% Confidence Interval); unit: Days to event
Arm/Group | Experimental | Control
Number analyzed (Participants) | 96 | 92
Days to event | 642 [370 to 1054] | 613 [226 to NA] — the upper confidence limit is not estimable due to insufficient number of participants with events after reaching the median time point
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.812, Log Rank

34. Secondary Outcome: The Percent of Participants With a Serum Creatinine of More Than 3 mg/dL.
Description: Serum creatinine (mg/dL) is used to measure kidney function. A normal result is 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women. Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys. This endpoint is ascertaining slow graft function in the immediate days post-transplant. A participant was considered to have met this endpoint if their day 5 serum creatinine was greater than 3 mg/dL.
Time Frame: Day 5 post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants who did not experience delayed graft function and with available serum creatinine data at day 5 post-transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 70
percentage of participants | 47.4 [36.0 to 59.1] | 42.9 [31.1 to 55.3]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.576, Chi-squared

35. Secondary Outcome: Creatinine Reduction Ratio (CRR), Defined as the First Creatinine on Day 2 Divided by he First Creatinine After Surgery
Description: Serum creatinine (mg/dL) is used to measure kidney function. A normal result is 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women. Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys. CRR was calculated as the day 1 post-transplant creatinine value minus the day 2 creatinine value divided by the day 1 creatinine value and multiplied by 100, resulting in a percentage. Higher numbers indicate a greater reduction in serum creatinine and, thus, potentially better kidney function.
Time Frame: Day 2 post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants who did not experience delayed graft function and with available serum creatinine data on days 1 and 2 post-transplant.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Experimental | Control
Number analyzed (Participants) | 77 | 70
Percentage | 24.28 (22.60) | 20.97 (16.64)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.311, t-test, 2 sided

36. Secondary Outcome: Creatinine Reduction Ratio (CRR), Defined as the First Creatinine on Day 5 Divided by the First Creatinine After Surgery.
Description: Serum creatinine (mg/dL) is used to measure kidney function. A normal result is 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women. Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys. CRR was calculated as the day 1 post-transplant creatinine value minus the day 5 creatinine value divided by the day 1 creatinine value and multiplied by 100, resulting in a percentage. Higher numbers indicate a greater reduction in serum creatinine and, thus, potentially better kidney function.
Time Frame: Day 5 post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants who did not experience delayed graft function and with available serum creatinine data on days 1 and 5 post-transplant.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 69
Percentage | 47.06 (28.86) | 43.37 (25.79)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.418, t-test, 2 sided

37. Secondary Outcome: The Percent of Participants Whose Day 5 Serum CRR Was Less Than 70%.
Description: Serum creatinine (mg/dL) is used to measure kidney function. A normal result is 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women. Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys. CRR was calculated as the day 1 post-transplant creatinine value minus the day 5 creatinine value divided by the day 1 creatinine value and multiplied by 100, resulting in a percentage. Higher numbers indicate a greater reduction in serum creatinine and, thus, potentially better kidney function. A participant was considered to have met this endpoint if their day 5 serum CRR was less than 70%.
Time Frame: Day 5 post-transplantation
Population: as for outcome 36
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 69
percentage of participants | 74.4 [63.2 to 83.6] | 88.4 [78.4 to 94.9]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.030, Chi-squared

38. Secondary Outcome: The Percent of Participants Whose Day 2 Serum CRR Was Less Than 30%.
Description: Serum creatinine (mg/dL) is used to measure kidney function. A normal result is 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women. Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys. CRR was calculated as the day 1 post-transplant creatinine value minus the day 2 creatinine value divided by the day 1 creatinine value and multiplied by 100, resulting in a percentage. Higher numbers indicate a greater reduction in serum creatinine and, thus, potentially better kidney function. A participant was considered to have met this endpoint if their day 2 serum CRR was less than 30%.
Time Frame: Day 2 post-transplantation
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 77 | 70
percentage of participants | 57.1 [45.4 to 68.4] | 68.6 [56.4 to 79.1]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.153, Chi-squared

39. Secondary Outcome: The Percent of Participants Who Need Dialysis After Week 1.
Description: Participants who needed dialysis after the first week post-transplant were considered to have met this endpoint.
Time Frame: 1 week to 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants who did not experience delayed graft function and with available data after week 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 78 | 71
percentage of participants | 9.0 [3.7 to 17.6] | 2.8 [0.3 to 9.8]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.171, Fisher Exact

40. Secondary Outcome: Percent of Participants With de Novo DSA.
Description: Donor specific antibody (DSA) can be formed post-transplant as part of the recipient's alloimmune response to the transplanted organ. DSA was determined by a central laboratory. Participants with newly developed DSA (i.e., de novo) following transplant were considered to have met this endpoint.
Time Frame: 24 months post-transplantation
Population: Intent-to-treat population included all transplanted and randomized participants who received the infliximab/placebo infusion, subset to participants who had available DSA data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 112 | 110
percentage of participants | 8.0 [3.7 to 14.7] | 3.6 [1.0 to 9.0]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.163, Chi-squared

41. Secondary Outcome: Percent of Participants With Any Infection Requiring Hospitalization or Resulting in Death.
Description: Participants were considered to have met this endpoint if they had an infection that required hospitalization or resulted in death.
Time Frame: 24 months post-transplantation
Population: Safety population included all participants who received at least a portion of the infliximab/placebo infusion. This population includes one participant in the Experimental group who received some of the infliximab infusion prior to the transplant procedure being aborted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 114 | 112
percentage of participants | 43.0 [33.7 to 52.6] | 39.3 [30.2 to 49.0]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.572, Chi-squared

42. Secondary Outcome: Percent of Participants With Mycobacterial or Fungal Infections
Description: Participants were considered to have met this endpoint if they had at least one mycobacterial of fungal infection.
Time Frame: 24 months post-transplantation
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 114 | 112
percentage of participants | 6.1 [2.5 to 12.2] | 6.3 [2.5 to 12.5]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.973, Chi-squared

43. Secondary Outcome: Percent of Participants With CMV Viremia That Require a Change in Immunosuppression or Anti-viral Treatment as Per Standard of Care at the Site
Description: Participants were considered to have met this endpoint if they had a reported case of CMV viremia that required a change in their existing immunosuppression or the use of anti-viral therapy.
Time Frame: 24 months post-transplantation
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 114 | 112
percentage of participants | 18.4 [11.8 to 26.8] | 11.6 [6.3 to 19.0]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.152, Chi-squared

44. Secondary Outcome: Percent of Participants With BK Viremia That Require a Change in Immunosuppression or Anti-viral Treatment as Per Standard of Care at the Site.
Description: Participants were considered to have met this endpoint if they had a reported case of BK viremia that required a change in their existing immunosuppression or the use of anti-viral therapy.
Time Frame: 24 months post-transplantation
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 114 | 112
Percent of participants | 28.9 [20.8 to 38.2] | 13.4 [7.7 to 21.1]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.004, Chi-squared

45. Secondary Outcome: Percent of Participants With Malignancy.
Description: Participants were considered to have met this endpoint if they had a reported case of malignancy.
Time Frame: 24 months post-transplantation
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 114 | 112
Percent of Participants | 1.8 [0.2 to 6.2] | 0.9 [0.0 to 4.9]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p > 0.999, Fisher Exact

46. Secondary Outcome: Percent of Participants With Impaired Wound Healing Manifested by Wound Dehiscence, Wound Infection, or Hernia at the Site of the Transplant Incision
Description: Participants were considered to have met this endpoint if they had a reported case of impaired wound healing at the site of the transplant incision manifested by one wound dehiscence, wound infection, or hernia.
Time Frame: 24 months post-transplantation
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 114 | 112
Percent of participants | 7.9 [3.7 to 14.5] | 11.6 [6.3 to 19.0]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.347, Chi-squared

ADVERSE EVENTS:
Time Frame: From initiation of the investigational treatment through end of study, up to 60 months post-transplant
Description: Events grade 2 or higher were collected before protocol v4.0. Starting with protocol v4.0, non-serious AE grade 3 or higher were collected. All adverse events meeting serious criteria regardless of severity grade were collected. AE/SAE information was recorded by sites on electronic case report form. SAEs included death, life-threatening events, hospitalization (or prolongation), inability to conduct normal life functions, birth defect, or condition requiring intervention to prevent these items.
Groups:
- Experimental: The experimental group received rabbit anti-thymocyte globulin (rATG, Thymoglobulin) co-administered with anti-TNFa (infliximab/Remicade") followed by maintenance therapy with tacrolimus, either Mycophenolate Mofetil/MMF or Mycophenolate Acid/MPA (or their generic equivalents) and prednisone. This group includes one subject who was randomized to the infliximab/Remicade" arm and received a partial infusion of infliximab/Remicade" prior to the transplant procedure being aborted.
- Control: The control group received rabbit anti-thymocyte globulin (rATG, Thymoglobulin) plus placebo (sterile normal saline) induction followed by maintenance therapy with tacrolimus, either Mycophenolate Mofetil/MMF or Mycophenolate Acid/MPA (or their generic equivalents) and prednisone,
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 3/114 | 5/112
Serious Adverse Events (participants affected / at risk) | 87/114 | 82/112
Other Adverse Events (participants affected / at risk) | 44/114 | 41/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=114) | Control (N=112)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (6) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperparathyroidism tertiary (Endocrine disorders) | 0 (0) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 3 (3)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 4 (4) | 9 (9)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
BK virus infection (Infections and infestations) | 3 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (3) | 5 (5)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (2) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 1 (1)
Corona virus infection (Infections and infestations) | 4 (4) | 5 (5)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 2 (2)
Cytomegalovirus enteritis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 5 (5) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Parvovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Perinephric abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 7 (9)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Polyomavirus-associated nephropathy (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 3 (3) | 7 (8)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tick-borne fever (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (10) | 10 (13)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 8 (9) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delayed graft function (Injury, poisoning and procedural complications) | 8 (8) | 12 (12)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft loss (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Perinephric collection (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural persistent drain fluid (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal transplant torsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Donor specific antibody present (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4) | 4 (4)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Hypomania (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 7 (8)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Post procedural drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 3 (3)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 2 (2)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=114) | Control (N=112)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 8 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (1) | 2 (2)
BK virus infection (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Injection site infection (Infections and infestations) | 0 (0) | 1 (1)
Polyomavirus-associated nephropathy (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delayed graft function (Injury, poisoning and procedural complications) | 8 (8) | 6 (6)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (5) | 9 (10)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (12) | 8 (8)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney fibrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular atrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal vasculitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteral stent removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02495077/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02495077/SAP_001.pdf